CLINICAL TRIAL: NCT04361097
Title: Fecal Microbiota Transplantation as a Therapeutic Strategy in the Progression of Chronic Kidney Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario Dr. Jose E. Gonzalez (Other)
Responsible Party: Principal Investigator, Dr. Adrian Camacho-Ortiz, MD, Hospital Universitario Dr. Jose E. Gonzalez
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IF18-00003
Record Dates: First submitted 2020-04-22; First posted 2020-04-24 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Chronic Kidney Disease Due to Hypertension; Chronic Kidney Disease Due to Type 2 Diabetes Mellitus
Keywords: chronic kidney disease; fecal microbiota
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Intervention Model Description: Prospective, double blind, experimental
Who Masked: Participant, Care Provider, Investigator
Masking Description: Third party makes the aleatorization
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Faecal microbiota transplant (Experimental): This group will receive frozen capsules to be ingested orally constituted of TMF with a frequency of 15 capsules every 12hrs for 4 doses on days 1, 10 and 30 of the study. Each capsule should be ingested in a period no longer than 1 hour.
  Interventions: Biological: Faecal microbiota transplant
- Placebo (Placebo Comparator): This group will receive frozen capsules to be ingested orally placebo with a frequency of 15 capsules every 12hrs for 4 doses on days 1, 10 and 30 of the study. Each capsule should be ingested in a period no longer than 1 hour.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Faecal microbiota transplant — Both groups will receive frozen capsules to be ingested orally (constituted of TMF or placebo according to the randomization) with a frequency of 15 capsules every 12hrs for 4 doses on days 1, 10 and 30 of the study. Each capsule should be ingested in a period no longer than 1 hour.
  Arms: Faecal microbiota transplant
Biological: Placebo — Both groups will receive frozen capsules to be ingested orally (constituted of TMF or placebo according to the randomization) with a frequency of 15 capsules every 12hrs for 4 doses on days 1, 10 and 30 of the study. Each capsule should be ingested in a period no longer than 1 hour.
  Arms: Placebo

SUMMARY:
What the investigators want to achieve with the protocol is to identify the impact of intestinal microbiota transplantation on the progression of chronic kidney disease.

Hypothesis: Modification of intestinal microbioma of CKD patients by TMF decrease the progression of CKD Methodological design: Experimental, prospective, double-blind. Inclusion criteria: Being diagnosed with CKD and creatinine clearance less than 60 mL/minute secondary hypertension and/or diabetes and older than 18 years

DETAILED DESCRIPTION:
What the investigators want to achieve with the protocol is to identify that impact has transplantation intestinal microbiota on the progression of chronic kidney disease

A.-Hypothesis: Modification of intestinal microbioma of CKD patients by TMF decrease the progression of CKD.

B.-Specific objectives: Evaluate whether decreases TMF markers of inflammation in patients with CKD after being treated with TMF, evaluate the behavior in CKD progression markers in patients undergoing TMF, evaluate the change in bowel microbioma CKD patients before and after undergoing TMF.

C.-Methodological design: Experimental, prospective, double-blind.

D.-Type of study: Controlled clinical trial

E.- Population in study:

1. -Inclusion criteria: Being diagnosed with CKD and creatinine clearance less than 60 mL/minute secondary hypertension and/or diabetes, older than 18 years.
2. - Exclusion Criteria: Malignancies whose last treatment has been less than 5 years, he is receiving antibiotics for any reason during the month prior to enrollment, having received probiotics in the last 3 months, it has been diagnosed with Clostridium difficile infection in the last year, it has been previously subjected to TMF , exacerbations of submitting ERC during the 3 months prior or present at the time of enrollment.
3. -Criteria for elimination: Failure to comply in the structured patient monitoring, nondelivery of stool samples at set times, the patient decides to no longer participate in the study.

F.- Desing Description: After being selected and randomized patients who meet the criteria for inclusion and exclusion, they are assigned to a group to start treatment TMF (capsules intestinal microbiota frozen) or a group receive placebo capsules which shall consist of an excipient harmless to the body (capsules frozen saline), both will be developed in the service Infectología.

Both groups receive frozen for ingestion orally capsules (comprised of TMF or placebo according to the randomization) with a frequency of 15 capsules each 12hrs for 4 doses on days 1, 10 and 30 of the study. Each capsule must be ingested over a period no longer than 1 hour.

measurements characteristic factors of the progression of kidney disease day 0,10, 30, 60, 90, 120 and 180 be made consisting of:

* Proteins in urine 24 hours
* Creatinine clearance 24 hours
* CBC
* serum creatinine
* Urea Nitrogen
* Urea
* Glucose
* Uric acid
* IS
* venous gases

Blood samples were taken by puncture of peripheral vein by laboratory personnel to assess renal function, urine samples will be collected by the patient at home and transported to the laboratory, none of these samples will be used for genetic analysis , only samples of faeces they underwent genomic analysis, collection of stool samples will days 0, 5, 10 30, 90 and 180 (on 10, 30, 90 and 180 with a range of +/- 2 days).

adverse effects questionnaires on days 1, 5, 30 and 60 is performed and quality of life assessment on days 0, 10, 30, 90 and 180.

Monitoring will face on a weekly basis to register if they have submitted infections, adverse effects and whether changes have received treatment. Visits will be made in the epidemiology and the Regional Center for Kidney Diseases University Hospital

ELIGIBILITY:
Inclusion Criteria:

* Be diagnosed with CKD and creatinine clearance less than 60 ml / minute secondary to hypertension and / or diabetes.
* Age over 18 years

Exclusion Criteria:

* Malignant neoplasms whose last treatment was less than 5 years
* Having received antibiotics for any reason during the month prior to enrollment
* Have received probiotics in the last 3 months
* Have been diagnosed with Clostridium difficile infection in the last year
* Have been previously submitted to TMF
* Having presented ERC exacerbations during the 3 months prior or present at the time of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2018-08-07 (Actual); Primary Completion 2019-11-07 (Actual); Study Completion 2020-04-21 (Actual)

PRIMARY OUTCOMES:
Creatinine Clearance | 6 months
  Arrest CKD progression

SECONDARY OUTCOMES:
24-hour Urine Protein | 6 months
  Arrest CKD progression
Serum Creatinine | 6 months
  Arrest CKD progression
Hemoglobin | 6 months
  Arrest CKD progression
Hematocrit | 6 months
  Arrest CKD progression
Leukocytes | 6 months
  Arrest CKD progression
Neutrophils | 6 months
  Arrest CKD progression
Platelets | 6 months
  Arrest CKD progression
Glucose | 6 months
  Arrest CKD progression
Urea Nitrogen | 6 months
  Arrest CKD progression
Uric Acid | 6 months
  Arrest CKD progression
Albumin | 6 months
  Arrest CKD progression
Reactive Protein C | 6 months
  Arrest CKD progression
Chlorine | 6 months
  Arrest CKD progression
Sodium | 6 months
  Arrest CKD progression
Potassium | 6 months
  Arrest CKD progression
Phosphorous | 6 months
  Arrest CKD progression
pH Venous Gasometry | 6 months
  Arrest CKD progression
CO2 pressure venous | 6 months
  Arrest CKD progression
Venous Bicarbonate | 6 months
  Arrest CKD progression
Base Excess | 6 months
  Arrest CKD progression
Lactate | 6 months
  Arrest CKD progression

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Camacho-Ortiz, PhD, Principal Investigator — Hospital Universitario "Dr. Jose Eleuterio Gonzalez, UANL
Locations (1):
- Hospital Universitario José E. Gonzalez, Monterrey, Nuevo León, Mexico

REFERENCES:
- [Background] Choi HH, Cho YS. Fecal Microbiota Transplantation: Current Applications, Effectiveness, and Future Perspectives. Clin Endosc. 2016 May;49(3):257-65. doi: 10.5946/ce.2015.117. Epub 2016 Mar 9. PMID 26956193
- [Background] Cruz-Mora J, Martinez-Hernandez NE, Martin del Campo-Lopez F, Viramontes-Horner D, Vizmanos-Lamotte B, Munoz-Valle JF, Garcia-Garcia G, Parra-Rojas I, Castro-Alarcon N. Effects of a symbiotic on gut microbiota in Mexican patients with end-stage renal disease. J Ren Nutr. 2014 Sep;24(5):330-5. doi: 10.1053/j.jrn.2014.05.006. Epub 2014 Jul 22. PMID 25066654
- [Background] Felizardo RJ, Castoldi A, Andrade-Oliveira V, Camara NO. The microbiota and chronic kidney diseases: a double-edged sword. Clin Transl Immunology. 2016 Jun 10;5(6):e86. doi: 10.1038/cti.2016.36. eCollection 2016 Jun. PMID 27757226
- [Background] Guida B, Germano R, Trio R, Russo D, Memoli B, Grumetto L, Barbato F, Cataldi M. Effect of short-term synbiotic treatment on plasma p-cresol levels in patients with chronic renal failure: a randomized clinical trial. Nutr Metab Cardiovasc Dis. 2014 Sep;24(9):1043-9. doi: 10.1016/j.numecd.2014.04.007. Epub 2014 May 2. PMID 24929795
- [Background] Honda K, Littman DR. The microbiota in adaptive immune homeostasis and disease. Nature. 2016 Jul 7;535(7610):75-84. doi: 10.1038/nature18848. PMID 27383982
- [Background] Jha V, Garcia-Garcia G, Iseki K, Li Z, Naicker S, Plattner B, Saran R, Wang AY, Yang CW. Chronic kidney disease: global dimension and perspectives. Lancet. 2013 Jul 20;382(9888):260-72. doi: 10.1016/S0140-6736(13)60687-X. Epub 2013 May 31. PMID 23727169
- [Background] Kelly CR, Ihunnah C, Fischer M, Khoruts A, Surawicz C, Afzali A, Aroniadis O, Barto A, Borody T, Giovanelli A, Gordon S, Gluck M, Hohmann EL, Kao D, Kao JY, McQuillen DP, Mellow M, Rank KM, Rao K, Ray A, Schwartz MA, Singh N, Stollman N, Suskind DL, Vindigni SM, Youngster I, Brandt L. Fecal microbiota transplant for treatment of Clostridium difficile infection in immunocompromised patients. Am J Gastroenterol. 2014 Jul;109(7):1065-71. doi: 10.1038/ajg.2014.133. Epub 2014 Jun 3. PMID 24890442
- [Background] Lin CJ, Wu V, Wu PC, Wu CJ. Meta-Analysis of the Associations of p-Cresyl Sulfate (PCS) and Indoxyl Sulfate (IS) with Cardiovascular Events and All-Cause Mortality in Patients with Chronic Renal Failure. PLoS One. 2015 Jul 14;10(7):e0132589. doi: 10.1371/journal.pone.0132589. eCollection 2015. PMID 26173073
- [Background] Marotz CA, Zarrinpar A. Treating Obesity and Metabolic Syndrome with Fecal Microbiota Transplantation. Yale J Biol Med. 2016 Sep 30;89(3):383-388. eCollection 2016 Sep. PMID 27698622
- [Background] Nallu A, Sharma S, Ramezani A, Muralidharan J, Raj D. Gut microbiome in chronic kidney disease: challenges and opportunities. Transl Res. 2017 Jan;179:24-37. doi: 10.1016/j.trsl.2016.04.007. Epub 2016 Apr 30. PMID 27187743
- [Background] Ramezani A, Massy ZA, Meijers B, Evenepoel P, Vanholder R, Raj DS. Role of the Gut Microbiome in Uremia: A Potential Therapeutic Target. Am J Kidney Dis. 2016 Mar;67(3):483-98. doi: 10.1053/j.ajkd.2015.09.027. Epub 2015 Nov 15. PMID 26590448
- [Background] Ranganathan N, Friedman EA, Tam P, Rao V, Ranganathan P, Dheer R. Probiotic dietary supplementation in patients with stage 3 and 4 chronic kidney disease: a 6-month pilot scale trial in Canada. Curr Med Res Opin. 2009 Aug;25(8):1919-30. doi: 10.1185/03007990903069249. PMID 19558344
- [Background] Rossi M, Johnson DW, Morrison M, Pascoe E, Coombes JS, Forbes JM, McWhinney BC, Ungerer JP, Dimeski G, Campbell KL. SYNbiotics Easing Renal failure by improving Gut microbiologY (SYNERGY): a protocol of placebo-controlled randomised cross-over trial. BMC Nephrol. 2014 Jul 4;15:106. doi: 10.1186/1471-2369-15-106. PMID 24996842
- [Background] Sabatino A, Regolisti G, Brusasco I, Cabassi A, Morabito S, Fiaccadori E. Alterations of intestinal barrier and microbiota in chronic kidney disease. Nephrol Dial Transplant. 2015 Jun;30(6):924-33. doi: 10.1093/ndt/gfu287. Epub 2014 Sep 4. PMID 25190600
- [Background] Vaziri ND, Wong J, Pahl M, Piceno YM, Yuan J, DeSantis TZ, Ni Z, Nguyen TH, Andersen GL. Chronic kidney disease alters intestinal microbial flora. Kidney Int. 2013 Feb;83(2):308-15. doi: 10.1038/ki.2012.345. Epub 2012 Sep 19. PMID 22992469

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-26): https://cdn.clinicaltrials.gov/large-docs/97/NCT04361097/Prot_SAP_000.pdf